CLINICAL TRIAL: NCT04580472
Title: Utility of Single-dose Oral Antibiotic Prophylaxis in Prevention of Surgical Site Infection in Dermatologic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Mariana Phillips, Section Chief of Dermatology & Mohs Surgery, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-19-482
Record Dates: First submitted 2020-09-03; First posted 2020-10-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cephalexin; Clindamycin

STUDY DESIGN:
Intervention Model Description: Patients meeting inclusion criteria will be assigned to one of three participant categories: 1) patients undergoing repair with skin flap or graft on the nose, 2) patients undergoing repair with skin graft, flap, or wedge resection on the ear, or 3) patients undergoing Mohs surgery with closure or partial closure or surgical excision on the lower extremity below the knee. Within each category, participants will be randomized into one of two groups: group one will receive a preoperative placebo pill and group two will receive preoperative antibiotic prophylaxis (either a single dose of Cephalexin 2g PO or single dose of Clindamycin hydrochloride 600 mg PO if allergy to penicillin or cephalosporin). These doses for cephalexin and clindamycin hydrochloride are standard doses for adults. The administration time of the oral antibiotics (as well for placebo group) will be 5-15 minutes prior to surgery in the nose and ear group and 30 minutes prior incision in the leg group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be told if they are receiving the antibiotic or placebo. Dermatologic surgeons who are performing the surgery and assessing for surgical site infections will be blinded to which arm of the study the patient is randomized. In order to accomplish this, study nurses will be responsible for randomizing each participant and will administer the antibiotic or placebo to each participant after each patient has consented and after the dermatologic surgeon has placed the order for "cephalexin/placebo" or "clindamycin/placebo" (based on patient's allergies) in the electronic medical record.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Placebo - leg (Placebo Comparator): If randomized to placebo group, 4 placebo capsules will be administered PO 30 minutes prior to incision in the leg group.
  Interventions: Other: Placebo capsules
- Antibiotic- leg (Experimental): The administration time of the oral antibiotics will be 30 minutes prior to incision in the leg group. 4-500 mg capsules of cephalexin will be administered to the patient. If there is concern for previous allergy to cephalexin, 4-150 mg capsules of clindamycin hydrochloride will be administered
  Interventions: Drug: Cephalexin
- Placebo- nose (Placebo Comparator): If randomized to placebo group, 4 placebo capsules will be administered PO 5-15 minutes prior to surgery on the nose.
  Interventions: Other: Placebo capsules
- Antibiotic- nose (Experimental): The administration time of the oral antibiotics will be 5-15 minutes prior to surgery on the nose. 4-500 mg capsules of cephalexin will be administered to the patient. If there is concern for previous allergy to cephalexin, 4-150 mg capsules of clindamycin hydrochloride will be administered PO.
  Interventions: Drug: Cephalexin
- Placebo- ear (Placebo Comparator): If randomized to placebo group, 4 placebo capsules will be administered PO 5-15 minutes prior to surgery on the ear.
  Interventions: Other: Placebo capsules
- Antibiotic- ear (Experimental): The administration time of the oral antibiotics will be 5-15 minutes prior to surgery on the ear. 4-500 mg capsules of cephalexin will be administered to the patient. If there is concern for previous allergy to cephalexin, 4-150 mg capsules of clindamycin hydrochloride will be administered PO.
  Interventions: Drug: Cephalexin

INTERVENTIONS:
Drug: Cephalexin — If randomized to the antibiotic group, a single dose of cephalexin or clindamycin hydrochloride (if concern for previous allergy to Cephalexin) will be given prior to surgery.
  Other Names: Clindamycin hydrochloride
  Arms: Antibiotic- ear; Antibiotic- leg; Antibiotic- nose
Other: Placebo capsules — Patients will receive 4 placebo capsules prior to surgery if randomized to placebo group.
  Arms: Placebo - leg; Placebo- ear; Placebo- nose

SUMMARY:
The purpose of the study is to assess the effectiveness of a single dose of preoperative antibiotic in reducing surgical site infections in certain dermatological procedures. Patients will undergo surgical excision or Mohs surgery as is clinically indicated and part of usual care. The study will be a double blinded, placebo-controlled clinical trial. Patients meeting inclusion criteria will be assigned to one of three participant categories: 1) patients undergoing repair with skin flap or graft on the nose, 2) patients undergoing repair with skin graft, flap, or wedge resection on the ear, or 3) patients undergoing Mohs surgery with closure or partial closure or surgical excision on the lower extremity below the knee. Within each category, participants will be randomized into one of two groups: group one will receive a preoperative placebo pill and group two will receive preoperative antibiotic prophylaxis (either a single dose of Cephalexin 2g PO or single dose of Clindamycin hydrochloride 600 mg PO if allergy to penicillin or cephalosporin).

Patients will followed for 30 days +/- 7 after surgery to evaluate for any surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* presenting to Carilion Clinic Dermatology and Mohs surgery in Roanoke, VA at Riverside 1
* suspected to undergo a single-staged repair including a skin flap or graft on the nose
* OR suspected to undergo single-staged repair including a skin graft or flap or wedge resection 1 on the ear
* OR undergoing Mohs with closure or partial closure or surgical excision on the lower extremity below the knee

Exclusion Criteria:

* patients with intellectual or mental impairment affecting ability to give informed consent
* use of any antibiotic (other than intervention) within 48 hours of the surgery suspected infection at time of surgery
* inability to take cephalexin or clindamycin hydrochloride due to allergy or intolerance current inflammatory skin disease affecting the surgical site
* Patients undergoing concurrent surgery to oral or nasal mucosa
* Patients who have had a recent prosthetic joint surgery within two years and have been told they require antibiotic prophylaxis.
* Patients who are currently pregnant, concerned they could be pregnant, actively trying to conceive, or missed last menstrual period that is not explainable by a birth control method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Development of surgical site infection within 30 days of surgery | 30 days
  Rate of surgical site infection occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Phillips, MD, Principal Investigator — Carilion Clinic Dermatology and Mohs Surgery
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT04580472/ICF_000.pdf